CLINICAL TRIAL: NCT00607607
Title: A Phase 2 Study of Oral MKC-1 Administered Twice Daily for 14 Consecutive Days Every 4 Weeks in Patients With Recurrent or Resistant Epithelial Ovarian Cancer or Advanced Endometrial Cancer
Brief Title: A Phase 2 Study of Oral MKC-1 in Patients With Ovarian or Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Carolyn Sidor, MD, MBA, EntreMed, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-103
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Ovarian Cancer; Endometrial Cancer
Keywords: ovarian cancer; endometrial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Ovarian Cancer Patients
  Interventions: Drug: MKC-1
- B (Experimental): Endometrial Cancer Patients
  Interventions: Drug: MKC-1

INTERVENTIONS:
Drug: MKC-1 — capsules, provided 125 mg/m2 BID x 14 days in 28 day cycles

SUMMARY:
Patients will be treated with MKC-1, twice daily for 14 consecutive days every four weeks (a cycle of MKC-1 chemotherapy), until disease progression or unacceptable toxicities. Patients will be stratified to Arm A (ovarian cancer) or Arm B (endometrial cancer), and will receive identical treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent (and HIPAA authorization for release of protected health information, as applicable) prior to any study related assessments.
2. Histologically confirmed epithelial ovarian cancer, primary peritoneal carcinomatosis, fallopian tube cancers, or endometrial cancer.
3. Age > 18 years at the time of consent.
4. Arm A: Ovarian Cancer Patients:

   * Must have failed at least one prior platinum based and one taxane based chemotherapeutic regimen. [Platinum failure is defined as platinum-refractory (progression while receiving a platinum-containing regimen) or platinum-resistant (disease progression within 6 months from completion of platinum containing regimen)].
   * Have measurable disease according to RECIST or CA 125 criteria according to GCIG (CA-125 value of > 2 xULN).
   * Have no more than 3 prior regimens for their disease.

   Arm B: Endometrial Cancer Patients:
   * Have no more than 3 prior regimens for their disease
   * Have measurable disease according to RECIST.
5. ECOG performance status of 0, 1, or 2.
6. The following laboratory results, within 10 days of MKC-1 administration:

   * Hemoglobin greater than or equal to 90 g/L (9 g/dL)
   * Absolute neutrophil count greater than or equal to 1.5 x 109/L
   * Platelet count greater than or equal to 100 x 109/L
   * Serum creatinine less than or equal to 1.5 x ULN (upper limit of normal)
   * AST less than or equal to 2.5 x ULN
   * Serum Albumin greater than or equal to 30 g/L (3.0 g/dL)
   * Total bilirubin less than or equal to ULN

Exclusion Criteria:

1. Administration of cancer specific therapy within the following periods prior to study drug initiation:

   * chemotherapy less than 3 weeks prior;
   * hormonal therapy less than one week prior;
   * radiation therapy less than 2 weeks prior.
2. Requirement for paracentesis > 2 liters/week.
3. Pregnant or breast-feeding women. Female patients must be postmenopausal, surgically sterile, or they must agree to use a physical method of contraception. Female patient with childbearing potential must have a negative pregnancy test within 10 days before the first MKC-1 administration.
4. Known CNS metastases unless treated, clinically stable, and not requiring steroids.
5. Clinical evidence of significant bowel obstruction, active uncontrolled malabsorption syndromes, or a history of total gastrectomy.
6. Uncontrolled hypercalcemia (serum calcium-corrected > 3 mmol/L [12 mg/dL]).
7. Serious cardiac condition (Class III/IV congestive heart failure according to New York Heart Association classification); documented acute myocardial infarction within the previous 6 months.
8. Any medical conditions that, in the investigator's opinion, would impose excessive risk to the patient. These include: infection requiring parenteral or oral anti-infective treatment, any altered mental status, or any psychiatric condition that would interfere with the understanding of the informed consent.
9. Patients with previous malignancies unless free of recurrence for at least 5 years except cured basal cell carcinoma of the skin or carcinoma-in-situ of the uterine cervix.
10. Treatment with antiretroviral therapy metabolized through CYP3A4 (including indinavir, nelfinavir, ritonavir and saquinavir).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Tumor response rate (based on tumor measurements according to the RECIST criteria) or CA-125 | Every 4 to 8 weeks

SECONDARY OUTCOMES:
Time to progression | Time of progression
Adverse events spontaneously declared by the patients or noted during physical examination and laboratory tests. | As reported

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (6):
- Canada (6):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec